CLINICAL TRIAL: NCT02334072
Title: The Effects of Different Airway Devices on Middle Ear Pressure in Pediatric Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Adiyaman University Research Hospital (Other)
Responsible Party: Principal Investigator, Dr. Ülkü Sabuncu, Dr, Adiyaman University Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Adiyaman/LMA-MEP
Record Dates: First submitted 2015-01-05; First posted 2015-01-08 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Local Pressure Effects; Simple Ear

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Classical (Experimental): Laryngeal mask airway (LMA) is manufactured from medical grade silicone rubber and is reusable. It consists of 3 main components: An airway tube, inflatable mask and mask inflation line. The airway tube is slightly curved to match the oropharyngeal anatomy, semirigid to facilitate atraumatic insertion and semitransparent, so that condensation and regurgitated material is visible. The distal aperture of the airway tube opens into the lumen of an inflatable mask and is protected by two flexible vertical rubber bars, called mask aperture bars, to prevent the epiglottis from entering and obstructing the airway. The laryngeal mask classical application will be done following anesthesia induction.
  Interventions: Device: Laryngeal mask classical application
- I-Gel (Experimental): I-Gel LMA is anatomically designed mask made of a gel-like thermoplastic elastomer. It has a drain tube for gastric aspiration. I-gel laryngeal mask application will be done following anesthesia induction.
  Interventions: Device: I-gel laryngeal mask application
- Cobra (Experimental): Cobra LMA consists of a translucent silicone airway tube with an inflatable cuff sited approximately two-thirds of the way to the tip, a 15-mm standard adapter and an expanded distal end with a smooth posterior surface. The cuff forms a seal in the upper pharynx and the distal end sits in the laryngopharynx. The distal grill is designed to sit over the laryngeal inlet.Cobra laryngeal mask application will be done following induction of anesthesia
  Interventions: Device: Cobra laryngeal mask application
- Supreme (Experimental): The Supreme LMA is a single-use polyvinyl chloride supraglottic device. High oropharyngeal leak pressures are important as they indicate airway protection, feasibility of positive pressure ventilation and likelihood of successful LMA placement.Supreme laryngeal mask application will be done following induction of anesthesia and anesthesia.
  Interventions: Device: Supreme laryngeal mask application
- Proseal (Experimental): The ProSeal LMA is the most complex of the specialized laryngeal mask devices.The primary design goal was to construct a laryngeal mask with improved ventilatory characteristics that also offered protection against regurgitation and gastric insufflation. The principal new features are a modified cuff and a drain tube.Proseal laryngeal mask application will be done following induction of anesthesia and anesthesia.
  Interventions: Device: Proseal laryngeal mask application

INTERVENTIONS:
Device: Laryngeal mask classical application — Laryngeal mask classical application will be done following induction of anesthesia and anesthesia will be conducted by this device.
  Arms: Classical
Device: I-gel laryngeal mask application — I-gel laryngeal mask application will be done following induction of anesthesia and anesthesia will be conducted by this device.
  Arms: I-Gel
Device: Cobra laryngeal mask application — Cobra laryngeal mask application will be done following induction of anesthesia and anesthesia will be conducted by this device.
  Arms: Cobra
Device: Supreme laryngeal mask application — Supreme laryngeal mask application will be done following induction of anesthesia and anesthesia will be conducted by this device.
  Arms: Supreme
Device: Proseal laryngeal mask application — Proseal laryngeal mask application will be done following induction of anesthesia and anesthesia will be conducted by this device.
  Arms: Proseal

SUMMARY:
Even though the effects of anesthetic agents both inhalation and intravenous have been well described, the effect of laryngeal mask airways haven't. The purpose of the study is to determine the effects of different types of laryngeal mask airways on middle ear pressure.

DETAILED DESCRIPTION:
All the patients in each group of laryngeal mask airway will contain 20 patients. In all groups middle ear pressures will be measured, in both right and left ear, preoperatively, after induction of anesthesia, insertion of laryngeal mask and in 1st., 5th., 10th. minutes and every 5 minutes perioperatively and recorded. Also the heart rates,arterial oxygen saturation (SaO2), airway pressures and end-tidal carbon dioxide values will be recorded before and following induction of anesthesia and in 1st., 5th., 10th. minutes and every five minutes perioperatively. Patients will be followed during the hospital stay for any complications.In all groups premedication will be done with midazolam. Anesthesia will be inducted with propofol and fentanyl; and maintained with sevoflurane-air combination.

ELIGIBILITY:
Inclusion Criteria:

* Elective patients undergoing subumbilical surgery under general anesthesia

Exclusion Criteria:

* Emergency conditions
* Rejection of patient approval
* Tympanic membrane perforation history
* Anticipated difficult airway
* Contraindications for LMA application

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-08 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Middle ear pressure changes after the device application (MEP) | Perioperative

SECONDARY OUTCOMES:
Composite Hemodynamics | Perioperative
  Heart rate,arterial blood pressure, haemoglobin saturation rate

CONTACTS AND LOCATIONS:
Overall Officials: Ruslan Abdullayev, Study Director — Adiyaman University Research Hospital
Locations (1):
- Adiyaman University Research Hospital, Adıyaman, Turkey (Türkiye)